CLINICAL TRIAL: NCT05008796
Title: Correlation Between PD-L1 Expression on Circulating Tumor Cells and Outcomes in Head and Neck Cancer Patients Treating With Curative Concurrent Chemo-radiotherapy
Brief Title: PD-L1 Expression on CTCs in HNSCC Patients Underwent Curative CCRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002049B0
Record Dates: First submitted 2021-08-12; First posted 2021-08-17 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Circulating Tumor Cell
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) is the 4th highest incidence of cancer and 6th of cancer death of the males in Taiwan. Because the patients were mainly middle-aged male, the disease eventually resulted in a huge loss of labor force, productivity and a huge burden of family supports and medicinal costs. Unfortunately, the incidence and death of HNSCC seemed to be increasing in Taiwan. Currently, the primary treatments of HNSCC are mainly surgery, radiotherapy, chemotherapy or targeted therapy or concurrent chemoradiotherapy. Immune checkpoint inhibitors become an emerging treatment in recent days. However, how to select adequate patient by using biomarkers remains an unsolved problem. Therefore, investigator have developed a new method for isolation and detection of circulating tumor cells (CTCs) in HNSCC patients. Moreover, the expression of immune markers (such as PD-L1, PD-L2, PD-1) on CTCs or immune cells might be a good target to study. Investigator's preliminary data found CTCs and circulating cancer stem-like cells but not PD-1 expression levels on peripheral T cells in patients with recurrence or metastasis HNSCC did not associated with overall survival. Therefore, investigators are wondering if PD-L1 more specific due to it expression on cancer cells. Therefore, in the 3-year project, investigators will utilize developing device and protocol in first year and then enroll 40 freshly diagnosed participants with head and neck cancer at stage III-IV with intent to receive curative concurrent chemo-radiotherapy (CCRT), and then analyze CTCs, PD-L1 expression levels on CTCs. Blood sample will be taken before, during (definition: 3-6 weeks after start RT) and after (definition: 4 +/-2 weeks after complete CCRT) completion of CCRT. Investigators will also enroll 10 health participants and taking blood sample for 3 times and follow up. Further statistical tests with clinical conditions (disease status, treatment effects, progression or distant metastasis and death) will be performed to elucidate their clinical significance. Hopefully, investigators will clarify the correlation between clinical outcomes and expression of PD-L1 on CTCs in head and neck patients. This could be a new biomarker for clinical cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck squamous cell carcinoma with age at diagnosis ≥ 20 years
* Stage III-IV according to AJCC 8th ed.
* Intent to receive curative concurrent chemoradiotherapy (CCRT)
* 10 healthy donors without any cancer diagnosis within 5 years

Exclusion Criteria:

* P16 positive oropharyngeal cancer
* Non-Platinum based CCRT
* Previous diagnosed with cancer within 3 years
* Synchronous cancer
* Poor compliance, cannot cooperate for blood sampling for CTCs isolation as time schedule or clinical treatment or follow-up

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stage III-IV head and neck squamous cell carcinoma patients, except those with P16 positive oropharyngeal cancer patients, who are going to do curative platinum-based CCRT.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 1 year

SECONDARY OUTCOMES:
Loco-regional recurrence rate | 1 year
Distant metastasis rate | 1 year
overall survival rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No